CLINICAL TRIAL: NCT02231671
Title: A Phase 1, Open-Label Study of the Absorption, Metabolism, Excretion and Absolute Bioavailability of 14C-ALS-008176 in Healthy Male Subjects
Brief Title: A Phase 1, Open-Label Study of the Absorption, Metabolism, Excretion and Absolute Bioavailability of ALS-008176
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ALS-008176-504
Record Dates: First submitted 2014-08-29; First posted 2014-09-04 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Absolute Bioavilability (Experimental): Part 1 of this study is an absolute bioavailability study where the IV (intravenous) microtracer dose of ALS-008112 is administered 15-30 minutes after the oral dose to determine the bioavailability of the oral dose compared to the IV dose. The maximum microtracer IV dose administered in Part 1 of this study will not exceed a single dose of 100 μg [14C]-ALS-008112 containing NMT (not more than) 37.0 kBq (1000 nCi) 14C. Based upon previous clinical observations, it is anticipated that the single oral dose and IV microdose to be utilised in Part 1 will provide acceptable PK data and will be safe and well tolerated.
  Interventions: Drug: ALS-008176; Drug: ALS-008112
- Part 2: Mass Balance (Experimental): Part 2 of this study is an absorption, metabolism and excretion study, for which a single 375 mg [14C]-ALS-008176 (containing NMT 6.85 MBq (megabecquerel) (185 μCi) 14C) dose has been selected for evaluation based upon data from prior studies. Based upon previous clinical observations, it is anticipated that the dose to be utilised in Part 2 will provide acceptable PK data, will be safe and well tolerated and is within the therapeutic range.
  Interventions: Drug: ALS-008176

INTERVENTIONS:
Drug: ALS-008176
Drug: ALS-008112
  Arms: Part 1: Absolute Bioavilability

SUMMARY:
The purpose of this study is to see how ALS-008176 is taken up, broken down, and removed from the body.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0 to 32.0 kg/m2 (inclusive) and a total body weight >50 kg

Exclusion Criteria:

* Creatinine clearance as calculated by the Cockroft-Gault formula of less than 60 mL/min
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator or the sponsor medical monitor. Reticulocyte count, haemoglobin and platelet counts must not be less than the lower limit of normal for the subject.
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory, GI, haematological, neurological, endocrinological, immunological, musculoskeletal disease or any uncontrolled medical illness (eg active infection) or psychiatric disorder, as judged by the investigator or medical monitor.
* Clinically significant abnormal electrocardiogram (ECG) findings

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08-31 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Absolute Bioavailability | Days 1-8
  Determination of the absolute bioavailability of ALS-008112
Mass Balance | Days 1 - 14
  Mass balance recovery of total radioactivity in urine, faeces, and urine and faeces combined: amount excreted (Ae) and Ae as a percentage of the administered dose (%Ae)

SECONDARY OUTCOMES:
Safety | Days 1-14
  Safety will be evaluated by recording adverse events, clinical laboratory results, vital signs, 12-lead ECGs, physical exams, etc.
To investigate the metabolic profile of [14C] - ALS-008176 | Days 1-14
  To investigate the metabolic profile of [14C] - ALS-008176 in plasma, urine and faeces following oral administration in healthy male subjects (Part 2 only)

CONTACTS AND LOCATIONS:
Overall Officials: Pui Leung, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom